CLINICAL TRIAL: NCT03366662
Title: The Effect of Frontal Electromyogram (F-EMG) Activity on the Entropy Index Behavior During General Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: lack of resources
Sponsor: Tampere University Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: R17108
Record Dates: First submitted 2017-12-01; First posted 2017-12-08 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia, General
Keywords: Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Monitoring of frontal electrical muscle activity — Continuous monitoring of frontal electrical muscle activity during general anesthesia simultaneous to burst suppression electroencephalogram

SUMMARY:
This study evaluates the effect of frontal EMG activity on Entropy index in burst suppression level of propofol anesthesia and surgery

DETAILED DESCRIPTION:
This is an academic observational study, where EEG is recorded during conventional propofol-remifentanil-rocuronium anesthesia and surgery in informed, consenting adults, during their surgical operations in Tampere University Hospital. The patients will be informed about the possibility to participate during their preoperative visit, and the approval will be asked on arrival in the day of surgery, before premedication.

The course of anesthesia will not be changed. The monitoring of the anesthetic state will be conventional: Heart rate, blood pressure, oxygen saturation of blood, Entropy Index, neuromuscular blockade will be monitored, as is the case in all surgical patients under general anesthesia in Tampere University Hospital. Any further monitoring will apply depending on the specific needs of the particular patient. Entropy Index data, EEG data and neuromuscular blockade data will be recorded on computer and analyzed later at GE Healthcare R&D Department, Helsinki, Finland, by Dr. Mika Särkelä. All data leaving Tampere University Hospital will be anonymized.

Anesthetic induction will be given in a conventional way (intravenous propofol and remifentanil, followed by intravenous rocuronium). EEG waveform is monitored with Entropy module. Neuromuscular blockade will be monitored with EMG-NMT module (GE-Healthcare). The data collection (Entropy, EEG, neuromuscular transmission (NMT) data) will last at least until skin incision.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled elective surgical operation under general anesthesia at Tampere University Hospital
* Written informed consent obtained

Exclusion Criteria:

* Subjects not giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients admitting to Tampere University Hospital for a scheduled surgical operation under general anesthesia
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Burst suppression electroencephalogram data without visible frontal electromyogram impact will be compared to burst suppression electroencephalogram data with visible frontal electromyogram impact on electroencephalogram signal | One day
  Visible EMG

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, PhD, Principal Investigator — Tampere University Hospital, Department of Anesthesia
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No